CLINICAL TRIAL: NCT05623592
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy of Methotrexate as Remission Maintenance Therapy After Remission-Induction Therapy With Tocilizumab and Glucocorticoids in Subjects With Giant Cell Arteritis
Brief Title: Methotrexate as Remission Maintenance Therapy After Remission-Induction With Tocilizumab and Glucocorticoids in Giant Cell Arteritis
Acronym: MTXinGCA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Valentin Schäfer, PD Dr. med. MuDr., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MED3-201802; EU-CT No: 2022-501058-12-00 (Other: EU Clinical Trials Register); DRKS-ID: DRKS00030571 (Other: German Clinical Trials Register)
Record Dates: First submitted 2022-11-08; First posted 2022-11-21 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Giant Cell Arteritis
Keywords: Giant cell arteritis; Methotrexate; Tocilizumab; Glucocorticoids; Remission maintenance; Vasculitis; Rheumatic disease; Ultrasound
MeSH Terms: conditions — Giant Cell Arteritis; Vasculitis; Rheumatic Diseases | interventions — Methotrexate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methotrexate (Experimental): The patient will be treated for 12 months weekly with methotrexate. Methotrexate will be provided at a dose of 17.5mg as a pre-filled syringe for self-injection. A dose reduction to 15 mg/week in case of intolerance, elevated liver enzymes >3x upper limit of normal or to 10 mg/week if glomerular filtration rate <50/min will be possible. If glomerular filtration rate <30/min, termination of treatment.
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Patients receive sodium chloride as a placebo subcutaneously. It will be administered in the form of a pre-filled syringe for self-injection once a week for 12 months.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Methotrexate — 17,5/15/10 mg Methotrexate subcutaneously
  Arms: Methotrexate
Drug: Sodium chloride — Sodium chloride subcutaneously
  Arms: Placebo

SUMMARY:
The standard treatment for Giant Cell arteritis (GCA) is Glucocorticoids(GC), even if GC-related adverse events are commonly occuring. Therefore, other practises for reducing relapses and cumulative GC-doses are needed. Currently, the Interleukin-6-inhibitor tocilizumab is used in combination with GC to achieve higher remission rates and lower cumulative GC-doses. The use of tocilizumab also has some disadvantages. One is the increased susceptibility to infections. On top of that, a long-term follow-up of the phase II study by Villiger et al. showed a 55% relapse-rate after discontinuation of intravenous tocilizumab after a median of five months.

Studies have also shown that methotrexate(MTX) in combination with GC was able to prevent relapses and reduce cumulative GC doses.

The aim of the study is to evaluate whether MTX is superior to placebo to prevent relapses in subjects with GCA after Remission-Induction Therapy with Glucocorticoids and Tocilizumab. Our hypothesis is that Methotrexate can maintain remission, once stable remission has been induced by GC and Tocilizumab and will prevent the occurrence of relapses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male or female, aged ≥18 years
* Written informed consent of the capable subject for voluntary participation in the study.
* Diagnosis of GCA as confirmed by the investigator fulfilment (also in retrospect) of the proposed extended 1990 classification criteria for GCA .
* Previous treatment with glucocorticoids and tocilizumab for new or relapsing GCA
* GCA patients who have been treated with tocilizumab and in whom discontinuation of tocilizumab therapy has been decided by the treating rheumatologist, within standard treatment at the department of rheumatology are eligible.
* total tocilizumab therapy should have been at least 6 months before inclusion.
* Patients should be in stable remission (defined as the absence of signs or symptoms of GCA and normal C-Reactive Protein (<1mg/dl), off glucocorticoids for at least 1 months at screening.
* Willing and able to inject methotrexate or placebo subcutaneously at randomization
* Male and female subjects agreeing to conduct efficient contraception (unless they have no childbearing potential)

Exclusion Criteria:

* Severe renal (glomerular filtration rate <30/min) failure
* Conditions other than GCA requiring continuous or intermittent treatment with oral or parenteral Glucocorticoids unless the last exposure to Glucocorticoids was >1 months before screening
* Other inflammatory rheumatic diseases (e.g. rheumatoid arthritis)
* Current treatment with any other conventional, biologic or targeted synthetic DMARD except tocilizumab
* Elevation of transaminases above three times the norm
* Simultaneous participation in another clinical trial, or participation in a clinical trial taking an investigational product, up to 30 days prior to participation in this clinical trial.
* Pregnant or breast feeding women
* Contraindications for therapy with Methotrexate, as indicated in the summary of product characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Time to relapse during the 12 months treatment period | 12 months

SECONDARY OUTCOMES:
Cumulative prednisone doses at months 6, 12 and 18 | 18 months
Number of relapses per patient during the 12 months treatment period | 12 months
Time to first, second and third relapse after randomization | 18 months
Percentage of patients with a relapse at month 6 and 18 after discontinuation of Tocilizumab | 18 months
Health-related quality of life: Short Form-36 | 18 months
  The possible score ranges from 0 to 100 points, where 0 points represent the greatest possible health limitation, while 100 points represent no health limitation at all
Self-reported fatigue : FACIT-Fatigue (Functional Assessment of Chronic Illness Therapy - Fatigue Scale) | 18 months
  The possible score ranges from 0 to 52 points. The higher this value, the better the quality of life.
Patient Global Assessment of disease activity (PGA) | 18 months
  The possible score ranges from 0 to 100 points, where 0 points represent the lowest disease activity and 100 the highest.
Patient Assessment of pain | 18 months
  The possible score ranges from 0 to 100 points, where 0 points represent the least pain intensity and 100 the most pain intensity
Investigator reported Evaluator Global Assessment of disease activity (EGA) | 18 months
  The possible score ranges from 0 to 100 points, where 0 points represent the lowest disease activity and 100 the highest.
Occurrence of symptoms and signs related to Giant cell arteritis | 18 months
Number of vasculitic vessels and change of intima-media-values of temporal and axillary arteries | 18 months
Prevalence of aortitis at baseline and month 12 and 18 in MRI | 18 months
Proportion of subjects with increased Erythrocyte Sedimentation Rate (>20mm/h) and C-Reactive Protein levels (> 10mg/L) | 18 months
Occurrence of adverse events and serious adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Valentin S. Schäfer, Dr. med., Principal Investigator — University Hospital of Bonn
Locations (1):
- Medical Clinic and Polyclinic III Internal medicine Oncology, Hematology University Hospital Bonn, Rheumatology and Clinical Immunology, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: We plan to share data, if an adequate proposal is submitted

REFERENCES:
- [Derived] Kreis L, Dejaco C, Schmidt WA, Nemeth R, Venhoff N, Schafer VS. The Meteoritics Trial: efficacy of methotrexate after remission-induction with tocilizumab and glucocorticoids in giant cell arteritis-study protocol for a randomized, double-blind, placebo-controlled, parallel-group phase II study. Trials. 2024 Jan 15;25(1):56. doi: 10.1186/s13063-024-07905-4. PMID 38225579